CLINICAL TRIAL: NCT01375751
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Tolerability and Efficacy of AMG 145 on LDL-C in Subject With Heterozygous Familial Hypercholesterolemia
Brief Title: Reduction of Low-Density Lipoprotein Cholesterol (LDL-C) With PCSK9 Inhibition in Heterozygous Familial Hypercholesterolemia Disorder Study
Acronym: RUTHERFORD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20090158
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Hypercholesterolemia, Familial
Keywords: Heterozygous Familial Hypercholesterolemia; Proprotein convertase subtilisin/kexin type 9 (PCSK9)
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia, Autosomal Dominant, 3 | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Placebo
- Evolocumab 350 mg (Experimental): Participants received 350 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 420 mg (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab 350 mg; Evolocumab 420 mg
Biological: Placebo — d by subcutaneous injection
  Arms: Placebo

SUMMARY:
The primary objective of this study was to evaluate the effect of 12 weeks of subcutaneous evolocumab (AMG 145), compared with placebo, on percent change from baseline in LDL-C in adults with heterozygous familial hypercholesterolemia (HeFH).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 75 years of age
* Diagnosis of heterozygous familial hypercholesterolemia by having met the diagnostic criteria outlined by the Simon Broome Register Group (Scientific Steering Committee 1991)
* On an approved statin, with or without ezetimibe, with stable dose(s) for at least 4 weeks
* Fasting Low-Density Lipoprotein Cholesterol (LDL-C) ≥ 100 mg/dL
* Fasting triglycerides ≤ 400 mg/dL

Exclusion Criteria:

* Homozygous familial hypercholesterolemia
* Low-Density Lipoprotein (LDL) or plasma apheresis within 12 months prior to randomization
* New York Heart Association (NYHA) III or IV heart failure, or known left ventricular ejection fraction < 30%
* Uncontrolled cardiac arrhythmia
* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months prior to randomization
* Type 1 diabetes; newly diagnosed or poorly controlled type 2 diabetes (HbA1c > 8.5%)
* Uncontrolled hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-08-02 (Actual); Primary Completion 2012-05-16 (Actual); Study Completion 2012-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Raal F, Scott R, Somaratne R, Bridges I, Li G, Wasserman SM, Stein EA. Low-density lipoprotein cholesterol-lowering effects of AMG 145, a monoclonal antibody to proprotein convertase subtilisin/kexin type 9 serine protease in patients with heterozygous familial hypercholesterolemia: the Reduction of LDL-C with PCSK9 Inhibition in Heterozygous Familial Hypercholesterolemia Disorder (RUTHERFORD) randomized trial. Circulation. 2012 Nov 13;126(20):2408-17. doi: 10.1161/CIRCULATIONAHA.112.144055. Epub 2012 Nov 5. PMID 23129602
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women 18 to to 75 years of age, with a diagnosis of heterozygous familial hypercholesterolemia, fasting low-density lipoprotein cholesterol (LDL-C) of ≥ 100 mg/dL, and fasting triglycerides ≤ 400 mg/dL were eligible for this study.
  The first patient was enrolled on 02 August 2011 and the last patient was enrolled on 20 February 2012.
Pre-assignment Details: Randomization was stratified on the basis of screening LDL-C level (< 130 mg/dL [3.4 mmol/L] or ≥ 130 mg/dL) and ezetimibe use at baseline (yes or no).
Period: Overall Study
Arm/Group | Placebo | Evolocumab 350 mg | Evolocumab 420 mg
Started | 56 | 56 | 56
Received Treatment | 56 | 55 | 56
Completed | 56 | 55 | 56
Not Completed | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (all randomized participants who received at least 1 dose of investigational product).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab 350 mg | Evolocumab 420 mg | Total
Number analyzed (Participants) | 56 | 55 | 56 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (11.3) | 47.6 (13.6) | 51.8 (13.0) | 49.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 25 | 21 | 78
  Male | 24 | 30 | 35 | 89
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 54 | 55 | 56 | 165
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 1 | 3 | 7
  Black or African American | 0 | 3 | 1 | 4
  White | 48 | 48 | 52 | 148
  Other | 4 | 3 | 0 | 7
  Mixed Race | 1 | 0 | 0 | 1
Stratification Factor: LDL-C Level [Number; unit: participants]
  < 130 mg/dL | 19 | 17 | 19 | 55
  ≥ 130 mg/dL | 37 | 38 | 37 | 112
Stratification Factor: Baseline Use Of Ezetimibe [Number; unit: participants]
  No | 20 | 19 | 20 | 59
  Yes | 36 | 36 | 36 | 108
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — LDL-C was measured using ultacentrifugation
  mg/dL | 160.8 (44.0) | 156.8 (46.1) | 149.5 (36.3) | 155.7 (42.3)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 182.7 (52.6) | 178.0 (51.7) | 171.0 (43.6) | 177.2 (49.4)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 125.2 (30.3) | 120.9 (29.3) | 119.3 (27.6) | 121.8 (29.0)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] | 4.895 (1.790) | 5.119 (1.923) | 4.857 (1.688) | 4.956 (1.795)
Apolipoprotein B/Apolipoprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] | 0.899 (0.277) | 0.901 (0.286) | 0.867 (0.264) | 0.899 (0.274)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: LDL-C was measured using ultracentrifugation.
Time Frame: Baseline and Week 12
Population: Full analysis set; Missing ultracentrifugation (UC) LDL-C data at Week 12 were imputed using last observation carried forward (LOCF) and calculated LDL-C.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 56 | 55 | 56
percent change | 1.12 (2.88) | -42.70 (2.93) | -55.24 (2.88)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 350 mg; The null hypothesis was that there was no mean difference in the percent change from baseline at Week 12 in LDL-C between evolocumab and placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -43.82, 95% CI 2-sided [-51.56 to -36.09], Standard Error of Mean 3.92 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo vs Evolocumab 420 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -56.36, 95% CI 2-sided [-64.06 to -48.67], Standard Error of Mean 3.90 — Placebo is the reference

2. Secondary Outcome: Absolute Change From Baseline in LDL-C at Week 12
Description: LDL-C was measured using ultracentrifugation.
Time Frame: Baseline and Week 12
Population: Full analysis set; LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 56 | 55 | 56
mg/dL | 4.2 (5.2) | -61.3 (5.4) | -80.5 (5.2)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -65.5, 95% CI 2-sided [-79.6 to -51.4], Standard Error of Mean 7.1 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -84.7, 95% CI 2-sided [-98.8 to -70.7], Standard Error of Mean 7.1 — Placebo is the reference

3. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 56 | 55 | 56
percent change | 2.48 (2.80) | -39.31 (2.86) | -50.98 (2.80)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -41.79, 95% CI 2-sided [-49.32 to -34.26], Standard Error of Mean 3.81 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -53.46, 95% CI 2-sided [-60.95 to -45.97], Standard Error of Mean 3.79 — Placebo is the reference

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; LOCF imputation was used
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 56 | 55 | 56
percent change | 2.86 (2.61) | -31.89 (2.66) | -43.34 (2.61)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -34.75, 95% CI 2-sided [-41.77 to -27.74], Standard Error of Mean 3.55 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -46.20, 95% CI 2-sided [-53.18 to -39.23], Standard Error of Mean 3.53 — Placebo is the reference

5. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; LOCF imputaton was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 56 | 55 | 56
percent change | 2.98 (2.73) | -33.69 (2.79) | -42.03 (2.73)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -36.66, 95% CI 2-sided [-44.01 to -29.32], Standard Error of Mean 3.72 — Placbo is the reference
Statistical Analysis 2: Comparison: Placebo vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -45.01, 95% CI 2-sided [-52.32 to -37.70], Standard Error of Mean 3.70 — Placebo is the reference

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B /Apolipoprotein A-1 Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 56 | 55 | 56
percent change | -4.10 (2.53) | -38.02 (2.58) | -48.74 (2.53)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -33.92, 95% CI 2-sided [-40.72 to -27.11], Standard Error of Mean 3.45 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; ANCOVA model includes treatment group and LDL-C level and baseline ezetimibe use as covariates; LS Mean Treatment Difference = -44.64, 95% CI 2-sided [-51.41 to -37.86], Standard Error of Mean 3.43 — Placebo is the reference

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Evolocumab 350 mg | Evolocumab 420 mg
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55 | 2/56
Other Adverse Events (participants affected / at risk) | 24/56 | 22/55 | 19/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | Evolocumab 350 mg (N=55) | Evolocumab 420 mg (N=56)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | Evolocumab 350 mg (N=55) | Evolocumab 420 mg (N=56)
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 1 | 1
Injection site pain (General disorders) | 1 | 5 | 2
Influenza (Infections and infestations) | 6 | 1 | 4
Nasopharyngitis (Infections and infestations) | 6 | 7 | 7
Sinusitis (Infections and infestations) | 1 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 5 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.